CLINICAL TRIAL: NCT05986045
Title: Establishing Natural History in an Advanced New CF Care Era
Brief Title: ENHANCE- Establishing Natural History in an Advanced New CF Care Era
Status: Not yet recruiting | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University Hospital of Limerick (Other); Cork University Hospital (Other); University College Hospital Galway (Other); Belfast Health and Social Care Trust (Other); NHS Lothian (Other Government); Alder Hey Children's NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Cardiff and Vale University Health Board (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other); Erasmus University Rotterdam (Other); Medizinische Hochschule Brandenburg Theodor Fontane (Other); Massachusetts General Hospital (Other); The Hospital for Sick Children (Other); Teagasc (Industry)
Responsible Party: Sponsor
Other Study IDs: ENHANCE
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: Newborn infants diagnosed with Cystic Fibrosis at newborn screening
  Interventions: Other: Quality of Life
- Cohort 2: Children with previous diagnosis of Cystic Fibrosis up to 5 years of age
  Interventions: Other: Quality of Life
- Control: Newborn infants without cystic fibrosis
  Interventions: Other: Quality of Life

INTERVENTIONS:
Other: Quality of Life — ENHANCE will collect natural history on all children with cystic fibrosis who are enrolled over a 5 year period

SUMMARY:
Measured outcomes for people with CF have improved dramatically over the last 20 years, even prior to the widespread introduction of cystic fibrosis transmembrane conductance regulator (CTFR) modulator treatments. The outlook for children with CF has improved significantly, with longer predicted survival and a lower likelihood of morbidity. This has accelerated recently. These changes have occurred within a short period of time, and there is much that we now do not understand about disease progression in children with CF and how this differs from children without CF. CF is an area which is fortunate to have well-developed and successful disease registries. CF registries have provided significant amounts of very useful data to guide improvement in treatment and outcomes over many decades. The power of registries comes from the collection of a well-defined set of important outcome measures in very large numbers of people over many years.

The outcome measures collected routinely in clinical care, which form part of the registries, are helpful in monitoring moderate-advances and symptomatic disease in people with CF. CF registries however do not tend to collect tomography(CT) scores, lung clearance index(LCI) or indeed repeated collection of biomarkers of disease activity such as sweat chloride which are increasingly relevant in an era of modulator therapies and reducing burden of symptomatic disease. We perceive an urgent need to complement registry data, cataloguing the changing natural history if early childhood CF by proactively collecting and curating sensitive, meaningful outcome data in a large cohort of children during this new era in Ireland and the UK.

The prevalence, presentation and natural history of disease manifestation of CF in young children will change significantly in the next decade with advances in the understanding and treatment of CF, including the use of therapies aimed at CFTR function. ENHANCE provides an opportunity to study these changes in real-time and in ways that are relevant to the CF community.

ELIGIBILITY:
Inclusion Criteria:

Children with CF attending one of the study centres and fulling one of the following:

* Newborn infant diagnoses with cystic fibrosis through newborn screening (excludes children with an uncertain diagnosis), or having 2 documented CF disease causing mutations.
* Children with CF (sweat chloride>60mmol/L or 2 CF disease causing mutations) aged 0-6 at study initiation
* Healthy control infants without CF

Exclusion Criteria:

* Children or their parents not willing or able to complete with study procedures or assessments.
* Co-morbidities in groups 1 and 2, unrelated to CF, that in the opinion of the investigator would substantially impact on study measurements and unduly affect the veracity of the outcome data, for example a diagnosis of inflammatory bowel disease or extreme prematurity.
* Children in the control group who are carriers of CFTR mutations or have chronic medical or GI/Liver conditions that in the opinion of the investigator would unduly affect the veracity of the outcome data.
* We will not exclude someone who subsequently joins a CF Investigational drug trial if they are happy to continue, but if possible, will time their annual ENHANCE data collection to fall outside the time period of any experimental study drug administration

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All participants with CF will be invited to participate in ENHANCE. We will ensure a presentative mix of mutation groups, sex, ages, ethnicity and location in all cohorts. We will target recruitment to cohorts 1 and 2 based on the following split of mutations: 50% F508del homozygous(FF), 20%heterozygous for F508del and a minimum function mutation(FMF), 20% heterozygous for F508del and a residual function/gating mutation or gating/other mutation and 10% with no currently treatable mutation(NON).
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
1. The incidence, prevalence and progression of structural lung disease | 60 Months
  Spirometry-controlled Computed Tomography
2. The long-term natural history of pulmonary function and ventilation homogeneity. | 60 Months
  Spirometry, Multiple Breath Washout
3. The incidence, prevalence and longitudinal progression of CF liver disease. | 60 Months
  Liver Ultrasound, Liver Function Tests
4. The prevalence, natural history and progression of exocrine pancreatic dysfunction | 60 Months
  Faecal Elastase Analysis
5. The longitudinal natural history of gastrointestinal symptoms, inflammation and the gut microbiome compared to a healthy control population | 60 Months
  Microbiome Analysis, Identification of inflammatory markers, Abdominal Symptom Scores
6. The longitudinal natural history of annual sweat chloride levels in infants and children of different ages, the influence of different treatments on this and its association with other outcomes | 60 Months
  Sweat chloride
7. The longitudinal natural history of mental health outcomes in children with CF compared to controls. | 60 Months
  Mental Health Quality Of Life Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Paul McNally, Principal Investigator — RCSI

IPD SHARING:
Plan to Share IPD: No